CLINICAL TRIAL: NCT06424223
Title: Tunnel Approach With Biphasic Calcium Phosphate and Acellular Dermal Matrix for Horizontal Ridge Augmentation.
Brief Title: Tunnel Access for Horizontal Alveolar Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Principal Investigator, University of Bari Aldo Moro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mini-invasiveRidgeAugmentation
Record Dates: First submitted 2024-05-02; First posted 2024-05-22 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Bone Atrophy, Alveolar; Bone Loss; Bone Resorption; Alveolar Bone Loss; Alveolar Bone Resorption
Keywords: Bone augmentation; Bone regeneration; Tissues augmentation; Ridge augmentation
MeSH Terms: conditions — Alveolar Bone Loss; Bone Diseases, Metabolic; Bone Resorption

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ridge augmentation (Experimental)
  Interventions: Procedure: Horizontal Ridge augmentation

INTERVENTIONS:
Procedure: Horizontal Ridge augmentation — A vertical full-thickness incision in the mesial aspect of the defect ridge.Microsurgery instruments is subsequently use to carefully elevate the full thickness of the mucosa.
  Extreme caution must be exercised during these maneuvers to avoid tissue perforation and to maintain the integrity of the periosteum.An dermal matrix is place into the tunnel. A pouch is create between the bone and the matrix and the Biphasic Calcium Phosphate is inserted into the tunnel until the desirable ridge dimensions are obtained. Primary closure of the vertical incisions was achieved with single interrupted sutures.

SUMMARY:
Minimally invasive procedures with the tunnel technique have been suggested to decrease patient post-operative discomfort and morbidity in oral bone regeneration. In the ridge augmentation tunnel technique, crestal incision and the release of the connective tissue are avoided in order to enhance the blood supply of the flap. This approach preserves the blood circulation and does not damage the periosteum The purpose of this study is to evaluate the clinical outcome of a minimally invasive technique for maxillofacial horizontal bone augmentation .

DETAILED DESCRIPTION:
Several techniques have been introduced to minimize the invasiveness involved in oral bone regeneration, to prevent the coronal advancement of the flap, which in turn reduces postoperative discomfort, swelling, complications, and mobility.

The tunnel technique involves making a vertical incision to access the bone defect and inserting the grafts. The significant benefit of this approach is that it may be closed without the need for periosteal incisions. Several tunnel techniques have been described in the literature using various biomaterials including bovine bone, synthetic bone, bovine bone block, allograft block bone, hidroxiapatite. This clinical study assesses the efficiency of a minimally invasive surgical technique for horizontal ridge augmentation using Biphasic Calcium Phosphate and Acellular Dermal Matrix.

This minimally invasive procedure aims to increase the horizontal volume of the edentulous ridge in both its bone component (through the use of Biphasic Calcium Phosphate) and its mucosal component (through the use of Acellular Dermal Matrix). Compared to other traditional techniques, this procedure, performed through a tunnel approach, would significantly reduce the invasiveness of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients had to be healthy according to System of the American Society of Anesthesiology (ASA) and aged 18 years or older

  * No general medical condition representing a contraindication to implant therapy
  * minimum 2 missing teeth in the maxilla or mandible from the canine to the second molar
  * No periodontal disease (periodontal probing depth <4 mm) or treated periodontitis
  * Good oral hygiene (full mouth plaque index<25%)
  * Adequate control of inflammation (full mouth bleeding on probing<25%)

Exclusion Criteria:

* smoking of more than 15 cigarettes a day • untreated periodontal disease
* pregnancy or breastfeeding at date of inclusion • acute infections
* keratinized mucosal tissue less than 2 mm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the achievement of an adequate thickness of the alveolar ridge ridge | 5 months
  Digital intraoral casts will be superimposed to value the gained thickness of the ridge.
  The assessment of volume increase in the alveolar ridge will be observed within the implant planning software by measuring the variation in the width of the edentulous ridge by matching three scans. The scans will be conducted at baseline (T0), five months after ridge augmentation (T1), and two months after implant insertion (T2). The matching will be performed using corresponding pairs of regions. The thickness of the alveolar ridges on the same cross-section at the level of the implants inserted will be measured in mm using the "distance" tool.

SECONDARY OUTCOMES:
Histological analysis of newly formed tissues. | 5 months
  A histological analysis will be conducted by the pathology laboratory of the Bari University Hospital on a bone biopsy taken at the same time as the implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Saverio Capodiferro, Study Director — University of Bari Aldo Moro; Professor Massimo Corsalini, Study Director — University of Bari Aldo Moro; Dr. D'Albis Giuseppe, Principal Investigator — University of Bari Aldo Moro
Locations (1):
- Giuseppe D'Albis, Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] D'Albis G, Forte M, Marini L, Mustakim KR, Pilloni A, Corsalini M, Capodiferro S. Horizontal Ridge Augmentation with Xenogeneic Bone, Hyaluronic Acid, and Dermal Matrix by Tunnel Technique: A Case Series. Dent J (Basel). 2026 Jan 4;14(1):25. doi: 10.3390/dj14010025. PMID 41590149